CLINICAL TRIAL: NCT04706572
Title: Golden Walk- A Wearable Technology Assessment and Biofeedback for Gait Rehabilitation in Parkinson's Disease Patients
Brief Title: Golden Walk as Measure of Gait Rehabilitation in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: University of Roma La Sapienza (Other); Università degli studi di Roma Foro Italico (Other)
Responsible Party: Principal Investigator, Antonella Peppe, Principal Investigator, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSantaLucia
Record Dates: First submitted 2019-10-08; First posted 2021-01-13 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Rehabilitation; Parkinson Disease; Locomotion Disorder, Neurologic; Rhythm; Abnormal
Keywords: Golden rhythm; Auditory cue; Parkinson's disease; Smartphone App; Gait analysis
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Golden Rhythm (Experimental): Administration of an external auditory cue based on Golden Rhythm
  Interventions: Other: Stimulation with external auditory bio-feedback
- Patients with Metronome (Placebo Comparator): Administration of an external auditory cue based on metronome binary rhythm
  Interventions: Other: Stimulation with external auditory bio-feedback

INTERVENTIONS:
Other: Stimulation with external auditory bio-feedback — Administration of an external cue based on a personalized Golden Ratio -rhythm or a metronome-rhythm through an ad-hoc App for Smartphone

SUMMARY:
Gait is specifically impaired in Parkinson's disease (PD). External auditory cue based on a binary rhythm tested in PD patients disappear when the stimulus is removed. Golden Ratio (GR)is intrinsic in the human gait, but in PD patients this GR has been found impaired. Aim of the study is the administration of an auditory external cue based on a personalized Golden Ratio-rhythm which could potentially assist people with PD to cope with the difficulties that they experience while walking, thus increasing their mobility and autonomy.

DETAILED DESCRIPTION:
Gait is specifically impaired in Parkinson's disease (PD). External auditory cue based on a binary rhythm has been successfully used in people with PD to improve their gait quality, but the beneficial effects disappear when the stimulus is removed. Recent evidences have shown that, in healthy subjects, the structure of walking relies on a number, called Golden Ratio (GR), based on a perfect proportion between different gait phases. While GR is known to be impaired in people with PD, there are few evidences that a GR-based auditory stimulus could support people with PD in counteracting gait alterations. As hypothesis, an auditory external cue based on a personalized GR-rhythm could assist people with PD to cope with the difficulties that they experience while walking, thus increasing their mobility and autonomy, and that the nature of this GR-rhythm allows to maintain the beneficial effects in time. Two personalized auditory rhythms (a binary rhythm and a GR-rhythm) will be alternatively administered to each participant (see diagram below). Patient-specific rhythms will administered by a user-friendly ad-hoc app for smartphone. Two assessments will be performed during these 24 weeks, to assess treatment efficacy. At the end of the 24th week, half of patients will continue with the GR-rhythm and, in a final assessment, we will see if the effect lasts over time.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD, as proposed by the Brain Bank Criteria for PD, since at least 5 years
* suffered from a rigid akinetic form of bilateral Parkinson's Disease (Hoehn and Yahr: 2-3), according to current criteria
* to be on stable treatment regimen for at least the 3 months before the recruitment
* Mini Mental State Examination score >24
* Do not vary the pharmacological treatment during the entire duration of the study
* Be tested in "ON" medication state

Exclusion Criteria:

* inability to stand or walk without aids or supports
* factors affecting gait such as hip replacement, musculoskeletal disorders, uncorrected vision or vestibular problems;
* inability to follow instructions;
* severe dysautonomia with marked hypotension, major depression, dementia, pregnancy, or cardiac pacemaker

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Golden Ratio-rhythm on Gait walking speed | 18 months
  Changes in walking speed between baseline and end of the study

SECONDARY OUTCOMES:
Efficacy of Golden Ratio-rhythm on stride lenght | 18 months
  Changes in stride length between baseline and end of the study and between more and less affected side
Efficacy of Golden Ratio-rhythm on toe clearance | 18 months
  Changes in toe clearance between baseline and end of the study and between more and less affected side
Efficacy of Golden Ratio-rhythm on hMaxMalleoli | 18 months
  Changes in maximum Malleoli heigth between baseline and end of the study and between more and less affected side
Efficacy of Golden Ratio-rhythm on stride to stance ratio | 18 months
  Changes in stride to stance ratio between baseline and end of the study and between more and less affected side

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Peppe, Principal Investigator — Fondazione Santa Lucia
Locations (1):
- IRCCS Santa Lucia, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No